CLINICAL TRIAL: NCT06986109
Title: Effect of Subanaesthetic Dose of Ketamine on Depth of Anaesthesia Consistency During Propofol Total Intravenous Anaesthesia Administered by Closed-loop Anaesthesia Delivery System in Adults Undergoing Elective Laparoscopic Surgery: a Randomised Controlled Study
Brief Title: Effect of Subanaesthetic Dose of Ketamine on Depth of Anaesthesia Consistency
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Nitin Sethi, DNB, Senior Consultant, Sir Ganga Ram Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: EC/03/25/2670
Record Dates: First submitted 2025-05-07; First posted 2025-05-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Anesthesia
Keywords: ketamine; propofol; Bi-spectral index; closed-loop anaesthesia delivery system
MeSH Terms: interventions — Ketamine; Propofol

STUDY DESIGN:
Intervention Model Description: One hundred and six participants (53/group) aged 18-65 years, ASA physical status I-II, of either sex, and undergoing elective laparosocpic surgery will be randomly divided into one of the two groups:
  Group I: Ketamine Group Prior to anaesthesia induction, a bolus dose of ketamine solution 0.05-ml/kg (concentration 5mg/ml) will be administered followed by continuous intraoperative ketamine infusion of 0.05-ml/kg /h along with automated propofol TIVA delivered using CLADS.
  Group II: Placebo Group Prior to anaesthesia induction, an equivalent volume bolus (0.05-ml/kg) of 0.9% normal saline will be administered and it will be followed by continuous intraoperative 0.9% normal saline infusion at 0.05-ml/kg /h along with automated propofol TIVA delivered using CLADS.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study drugs will be prepared by an independent investigator not involved in the conduct of case. Both the drugs will be administered as a bolus of 0.05-ml/kg followed by intraoperative infusion of 0.05-ml/kg/h. The investigator conducting the case and the patient will be blinded to the allocated intervention. The postoperative follow up of the patients will be done by an independent investigator who will be neither involved in the preparation of the study drugs or the conduct of the case.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine Group (Active Comparator): 100 mg of ketamine will be diluted in 20 ml of normal saline to make a ketamine concentration of 5mg/ml. Patients will receive a pre-induction bolus of ketamine solution at 0.05-ml/kg administered over 5-minutes and followed by maintenance infusion rate of 0.05-ml/kg /h throughout the duration of surgery. Anaesthesia induction and maintenance will be carried with propofol delivered and controlled by closed-loop anaesthesia delivery system (CLADS) a BIS-based feedback-loop automated anaesthesia delivery system. A target BIS value of '50' will be considered adequate for both induction and maintenance of anaesthesia.
  Interventions: Drug: Ketamine; Drug: Propofol
- Placebo Group (Active Comparator): 20-ml of normal saline will be taken and an equivalent volume will be used with a pre-induction bolus of 0.05-ml/kg administered over 5-minutes and followed by maintenance infusion rate of 0.05-ml/kg /h throughout the duration of surgery.Anaesthesia induction and maintenance will be carried with propofol delivered and controlled by closed-loop anaesthesia delivery system (CLADS) a BIS-based feedback-loop automated anaesthesia delivery system. A target BIS value of '50' will be considered adequate for both induction and maintenance of anaesthesia.
  Interventions: Drug: Propofol; Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Ketamine (concentration 5mg/ml) will be administered at 0.05-ml/kg over 5-minutes followed by continuous intraoperative ketamine infusion of 0.05-ml/kg /h.
  Arms: Ketamine Group
Drug: Propofol — Propofol administration rate will be controlled by a feedback loop facilitated by BIS monitoring using the conventional closed loop anaesthesia delivery system (CLADS). A BIS value of 50 will be used as the target point for induction and maintenance of anaesthesia.
Drug: Placebo — Normal saline bolus 0.05-ml/kg will be administered over 5-minutes and it will be followed by continuous intraoperative normal saline infusion at 0.05-ml/kg /h.
  Arms: Placebo Group

SUMMARY:
General Anaesthesia (GA) is a medical state of controlled unconsciousness that inhibits two dimensions of consciousness: the content and the level of consciousness. This state is achieved using various anaesthetic agents, with propofol being one of the most commonly used intravenous anaesthetics. Propofol is a gamma amino butyric acid (GABAA) receptor agonist, which affects both the content and level of anaesthesia.

In some cases, anaesthesiologists may choose to use an adjuvant drug, ketamine, in subanaesthetic doses during inhalation GA and propofol total intravenous anaesthesia (TIVA). Ketamine is an N-methyl D-aspartate (NMDA) receptor antagonist and is primarily employed for its analgesic properties. Unlike propofol, ketamine selectively affects only the content of consciousness.

The combination of propofol and ketamine appears to have dual effects on the dimensions of consciousness, with propofol affecting both content and level, and ketamine affecting only the content. This combination is likely to complement and improve the consistency of intraoperative anaesthesia depth.

However, studies have shown that the administration of ketamine with propofol TIVA, delivered through an automated anaesthesia delivery system using electroencephalogram (EEG) feedback signals from NeuroSENSE processed electroencephalogram (pEEG) monitor, has not demonstrated any significant benefit over the use of propofol alone.

Till now, the only study on propofol-ketamine co-administration used an uncommon NeuroSENSE pEEG monitoring system. Closed loop anaesthesia delivery system (CLADS) is a more precise, efficient, and robust mechanism to facilitate automated administration of propofol TIVA which employs the standard bispectral index (BIS) pEEG monitoring to control propofol TIVA delivery. Further evidence is desirable on depth of anaesthesia consistency when ketamine is co-administered with propofol TIVA, using CLADS This randomised controlled study will compare the effect of subanaesthetic dose of ketamine versus placebo (normal saline) on anaesthesia depth consistency in patients undergoing elective laparoscopic surgery under automated propofol TIVA using CLADS. All patients undergoing elective laparoscopic surgery will be screened, and those found eligible will be enrolled. Enrolled patients will receive CLADS-controlled propofol TIVA as standard. In intervention are, patients will additionally receive subanaesthetic dose of ketamine (0.25-mg/kg bolus followed by maintenance infusion 0.25-mg/kg/h) (ketamine group); in control arm, patients will receive normal saline as placebo in addition to propofol TIVA (placebo group).

DETAILED DESCRIPTION:
General Anaesthesia (GA) is a state of controlled unconsciousness that negatively affects a person's subjective experience or interaction with the external environment. GA inhibits two dimensions of consciousness: the content and the level of consciousness. The content of consciousness relates to a person's awareness or subjective experience, while the level of consciousness reflects the degree of wakefulness or arousal. Intravenous anaesthetics, such as propofol, which affect both the content and level of anaesthesia, are used for total intravenous anaesthesia (TIVA). Recently, there has been renewed interest in exploring the addition of anaesthetic adjuvants (ketamine, dexmedetomidine, lignocaine) that affect either the content or level of consciousness, or both, to propofol TIVA.

Propofol is a commonly used anaesthetic for administering TIVA. It acts on gamma-aminobutyric acid (GABAA) receptors in the brain, resulting in hyperpolarisation and inhibition of electrical activity in the neuronal circuits involving the cortex and the thalamus. It simultaneously activates the sleep-generating ventrolateral preoptic nuclei (VLPO) of the hypothalamus. The resultant effect is the depression of both the content and level of consciousness. Propofol causes a transition in electroencephalogram (EEG) waves from high-frequency, low-amplitude beta waves (13-25 Hz) and gamma oscillations (26-80 Hz) of the awake state to high-amplitude, slow delta waves (1-4 Hz) and alpha oscillations (9-12 Hz)

Ketamine is a dissociative anesthetic often used in subanesthetic doses alongside both inhalation general anesthesia (GA) and propofol total intravenous anesthesia (TIVA) due to its numerous benefits, including postoperative pain relief, reduced postoperative nausea and vomiting (PONV), and decreased shivering. It works by antagonizing the N-methyl D-aspartate (NMDA) receptor on the GABAergic inhibitory interneurons in the brain, leading to the disinhibition of excitatory or arousal-promoting neurons in the cortex. Additionally, it inhibits the VLPO nuclei of the hypothalamus. As the dose of ketamine increases, NMDA receptors on excitatory glutaminergic neurons are blocked, resulting in unconsciousness. Unlike propofol, ketamine's EEG signature is characterized by high-frequency, low-amplitude beta (13-25Hz) and gamma oscillations (25-32Hz). This unique mechanism of action, which selectively affects the content of consciousness, leads to a cataleptic state marked by dysphoria, hallucinations, and delirium.

The coadministration of propofol and ketamine has shown an additive effect on hypnosis. Additionally, evidence suggests that ketamine, like propofol, disrupts corticocortical neural activity affecting feedback neural circuits from the frontal to parietal cortex while preserving feedforward neural activity. The EEG signature of ketamine co-administered with propofol resembles that of propofol but with an augmented peak frequency of alpha wave oscillation. The propofol-ketamine combination, which appears to have both dual and solitary effects on dimensions of consciousness, is likely to improve intraoperative anesthesia depth consistency. Administering ketamine with propofol through an automated anesthesia delivery system using EEG feedback signals from the NeuroSENSE processed electroencephalogram (pEEG) monitor (NeuroWave Systems, Ohio, USA) (depth of hypnosis (DoH) index: WAVCNS index, value: '0' to '100') has demonstrated that a subanesthetic dose of ketamine maintains equivalent anesthesia depth consistency similar to when propofol is administered alone. Therefore, adding subanesthetic doses of ketamine to propofol TIVA neither compromises the automated system performance nor affects anesthesia depth consistency. Further evidence is desirable regarding propofol-ketamine TIVA administered by objective automated systems incorporating a feedback-loop mechanism using the bispectral index (BIS) (Medtronics, Minneapolis, USA) pEEG monitor (DoH index: BIS score, value: '0' to '100'), whose working algorithm differs from that of the WAVCNS index. One such automated system using the BIS pEEG monitor is the closed-loop anesthesia delivery system (CLADS). The use of CLADS in patients undergoing cardiac and non-cardiac surgery has demonstrated robust anesthesia depth consistency with propofol TIVA.

The investigators hypothesize that administration of subanaesthetic dose of ketamine will improve the intraoperative anaesthesia depth consistency as compared to placebo in adults undergoing elective laparoscopic surgery under automated propofol TIVA using CLADS.

The proposed randomised-controlled study aims to compare the effect of addition of subanaesthetic dose of ketamine versus placebo on anaesthesia depth consistency in patients undergoing elective laparoscopic surgery under automated propofol TIVA using CLADS.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I and II.
* Patients scheduled for elective laparoscopic surgery with estimated duration greater than 60-minutes.

Exclusion Criteria:

* Known uncontrolled cardiovascular disease (e.g., hypertension, systolic and diastolic dysfunction)
* Liver function abnormality (liver enzymes >2 times the normal range)
* Kidney function abnormality (serum creatinine >1.4 mg/dl)
* Known psychiatric or neurological disorder
* Known uncontrolled endocrine disorder (diabetes mellitus, hypothyroidism)
* Known allergy or hypersensitivity to the study drug
* Recent intake of sedative medication or anti-psychotic medication
* Substance abuse
* Anticipated need for postoperative ventilation
* Refusal to informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Anaesthesia depth consistency | During the surgical procedure, an average of 360 minutes
  It will be determined by the percentage of the anaesthesia time during which the BIS remained +/- 10 of the target BIS of 50

SECONDARY OUTCOMES:
Performance characteristic of propofol delivery system determined by calculating the median performance error (MDPE) | During the surgical procedure, an average of 360 minutes
  It will be determined using the Varvel criteria parameter :median performance error (MDPE). This parameter is calculated by the computer software which analyses the intraoperative BIS data. This parameter have no unit of measurement. It's just an abstract number. Higher the value means worse performance of propofol delivery system. It is not a scale.
Performance characteristic of propofol delivery system determined by calculating the median absolute performance error (MDAPE) | During the surgical procedure, an average of 360 minutes
  It will be determined using the Varvel criteria parameter: median absolute performance error (MDAPE).This parameter is calculated by the computer software which analyses the intraoperative BIS data. This parameter have no unit of measurement. Its just an abstract number.Higher the value means worse performance of propofol delivery system. It is not a scale.
Performance characteristic of propofol delivery system determined by calculating the wobble | During the surgical procedure, an average of 360 minutes
  It will be determined using the Varvel criteria parameter: wobble. This parameter is calculated by the computer software which analyses the intraoperative BIS data. This parameter have no unit of measurement. Its just a abstract number.Higher the value means worse performance of propofol delivery system. It is not a scale.
Performance characteristic of propofol delivery system determined by calculating the global score | During the surgical procedure, an average of 360 minutes
  It will be determined using the Varvel criteria parameter: global score. It is calculated using the formula Median absolute performance error + wobble / percentage of the anesthesia time during which the BIS remained +/- 10 of the target BIS of 50. This parameter have no unit of measurement. Its just a abstract number.Higher the value means worse performance of propofol delivery system. It is not a scale.
Propofol induction dose (mg/kg) | From start of propofol injection till target BIS value of '50' is achieved, an average of 5 minutes after beginning of anesthesia
  Dose of propofol required for induction of anaesthesia
Propofol maintenance dose (mg/kg/h) | From achieving target BIS value of '50' till skin closure, during the surgical procedure an average of 360 minutes
  Dose of propofol required for maintenance of anaesthesia
Intraoperative haemodynamic instability | From beginning of anaesthesia till 10 hours intraoperatively
  Episodes (frequency) of occurrence of hypotension, hypertension, bradycardia and tachycardia will be noted. Hypotension will be defined as decrease in systolic blood pressure below 90 mmHg or >20% fall from pre-induction baseline. Hypertension will be defined as increase in systolic blood pressure above 140 mmHg or > 20% change from the baseline. A heart rate <50 bpm will be defined as 'bradycardia'. 'Tachycardia' will be defined as heart rate >100-bpm.
Early recovery from anaesthesia (measured in minutes) | From end of anaesthesia till 20-minutes postoperatively
  Time taken by the patient to open his/her eyes after discontinuation of anaesthesia will be noted
Early recovery from anaesthesia (measured in minutes) | From end of anaesthesia till 20-minutes postoperatively
  Time taken for tracheal extubation after discontinuation of anaesthesia will be noted
Postoperative pain assesment | From the end of anaesthesia till 24-hours, postoperatively
  Will be assessed using the 11-point numeric rating scale (NRS) ('0': no pain to '10': worst possible pain).
Postoperative nausea and vomiting | From the end of anaesthesia till 24-hours, postoperatively
  Will be assessed using the 3-point PONV score ('0' = No emetic symptoms; '1' = nausea; '2' = vomiting)
Postoperative sedation | From the end of anaesthesia till 24-hours, postoperatively
  Modified observer's assessment of alertness/sedation scale (MOAA/S) will be used to assess postoperative sedation levels.26 The scale assesses the level of sedation with score range 0 to 5; score-0 means deeply sedated and score-5 means wide awake
Intraoperative awareness | From the end of anaesthesia till 48-hours, postoperatively
  Will be assessed using modified brice interview

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Sethi, DNB, Study Chair — Sir Ganga Ram Hospital, New Delhi, INDIA; Amitabh Dutta, MD, PGDHR, Study Director — Sir Ganga Ram Hospital, New Delhi, INDIA
Locations (1):
- Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi, India